CLINICAL TRIAL: NCT07309276
Title: A Phase II Clinical Study Evaluating the Combination Therapy of JS212 in Patients With Advanced Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS212-002-II-LC
Record Dates: First submitted 2025-12-15; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Advanced Lung Cancer
MeSH Terms: interventions — Injections; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Queue 1: JS212 + JS207 (Experimental): JS212 will be administered by intravenous infusion on Day 1 of each 21-day cycle.
  JS207 will be administered by intravenous infusion on Day 1 of each 21-day cycle.
  Interventions: Drug: JS212 for Injection; Drug: JS207 for Injection
- Queue 2: JS212 + Toripalimab (Experimental): JS212 will be administered by intravenous infusion on Day 1 of each 21-day cycle.
  Toripalimab will be administered by intravenous infusion on Day 1 of each 21-day cycle.
  Interventions: Drug: JS212 for Injection; Drug: Toripalimab
- Queue 3: JS212 + JS213 (Experimental): JS212 will be administered by intravenous infusion on Day 1 of each 21-day cycle.
  JS213 will be administered by intravenous infusion on Day 1 of each 21-day cycle.
  Interventions: Drug: JS212 for Injection; Drug: JS213 for Injection

INTERVENTIONS:
Drug: JS212 for Injection — Administered by intravenous infusion on Day 1 of each 21-day cycle.
Drug: JS207 for Injection — Administered by intravenous infusion on Day 1 of each 21-day cycle.
  Arms: Queue 1: JS212 + JS207
Drug: Toripalimab — Administered by intravenous infusion on Day 1 of each 21-day cycle.
  Arms: Queue 2: JS212 + Toripalimab
Drug: JS213 for Injection — Administered by intravenous infusion on Day 1 of each 21-day cycle.
  Arms: Queue 3: JS212 + JS213

SUMMARY:
This is a multicenter, open-label Phase II clinical study, with the main objective being to evaluate the investigator-assessed objective response rate of JS212 in combination therapy for advanced lung cancer. The aim is to explore the safety, tolerability, and preliminary efficacy of JS212 combined with JS207, Toripalimab, JS213 combined or not combined with chemotherapy.

DETAILED DESCRIPTION:
Part One:

The plan involves including patients with previously failed standard treatments in advanced NSCLC and ES-SCLC. It consists of two phases: safety introduction and clinical expansion, covering cohorts 1 to 3.

The safety introduction phase will explore the safety of the following combined regimens in the target population:

Queue 1: JS212 + JS207 Queue 2: JS212 + Toripalimab Queue 3: JS212 + JS213

Part Two:

It is planned to include lung cancer patients who have not received any systemic anti-tumor treatment for advanced NSCLC and ES-SCLC in the past. If the SMC decides to further combine chemotherapy, the safety introduction phase should also include to ensure the safety of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The age between 18 and 75 years old, and any gender.
2. Local advanced, metastatic or recurrent NSCLC.
3. ES-SCLC.
4. According to the Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), there must be at least one measurable lesion.
5. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
6. Expected survival period of ≥ 12 weeks.
7. The functions of important organs meet the requirements.
8. Female participants with reproductive capacity (WOCBP) who have sexual life with an unsterilized male partner and who have signed the informed consent must have a negative serum pregnancy test result within 7 days before the first administration, and must agree to take effective contraceptive measures from the time of signing the ICF until 7 months after the last administration of the study.
9. Unsterilized male participants who have sexual life with a fertile female partner must agree to use the effective contraceptive measures after signing the ICF until 4 months after the last administration of the study. During this period, sperm donation is prohibited.
10. The participants voluntarily participate in this study and sign the informed consent.

Exclusion Criteria:

1. Accompanying the following disease states:

1. Tumor histological or cytological pathological confirmation of combined large cell neuroendocrine carcinoma or sarcomatoid lesion, or NSCLC with small cell lung cancer component;
2. NSCLC patients with positive driver mutations;
3. Patients with known meningeal metastasis;
4. Patients with symptomatic brain metastases;
5. Uncontrolled pleural effusion, pericardial effusion, or recurrent ascites;
6. Unatable spinal cord compression;

2. Participants in Cohort 1 and Cohort 4 need to exclude any of the following conditions:

1. Within one month before the first use of the study drug, any clinically significant hemoptysis or tumor bleeding;
2. High bleeding risk; tumor invading important organs, high risks of perforation, esophageal-tracheal fistula, massive hemoptysis, etc.;
3. Obvious bleeding tendency or severe coagulation dysfunction history, etc;
4. Recent gastrointestinal perforation, gastrointestinal obstruction, trachea-esophageal fistula, abdominal fistula or intra-abdominal abscess, or currently having high-risk factors for hollow organ perforation/ fistula formation, or active inflammatory bowel disease, etc;
5. Presence of severe, non-healed or open wounds, active ulcers or untreated fractures;
6. Have poorly controlled hypertension;
7. Have used antiplatelet drugs or anticoagulant therapy within 14 days;
8. Have experienced a drug-related adverse event that led to permanent discontinuation of the medication during previous Bevacizumab and similar agent treatments;

3. Have received any of the following treatments:

1. Immune-mediated treatments (only for part Two);
2. Have received any investigational drug within 4 weeks or 5 half-lives before the first use of the study drug;
3. Have been enrolled in another clinical study;
4. Have undergone major surgery within 4 weeks;
5. Have received local small-scale radiotherapy within 14 days;

4.Have not recovered to ≤ CTCAE grade 1 toxicity or the level specified in the inclusion/exclusion criteria.

5.Have known allergies to any study treatment or its excipients or have experienced an allergic reaction.

6.Have experienced a drug-related AE that led to permanent discontinuation of the anti-PD-(L)1 antibody treatment.

7.Have any of the following cardiac examination results:

1. Long QT;
2. Left ventricular ejection fraction (LVEF) < 50%;

8.Have a history of diagnosed or suspected ILD, drug-induced pneumonia, or other severe lung diseases.

9.Have experienced a severe infection within 4 weeks.

10.Have a history of immunodeficiency, or have a history of organ transplantation and allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation.

11.Have active pulmonary tuberculosis infection.

12.Have active hepatitis.

13. Uncontrolled concurrent diseases.

14. Participants who were diagnosed with any other malignant tumor within 5 years.

15. Female participants who are pregnant, breastfeeding, or planning to become pregnant during the study period.

16. Other conditions for trial participation were not considered appropriate by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-11-11 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 6 years
  Objective response rate(ORR), assessed by BICR (RECIST v1.1)

SECONDARY OUTCOMES:
PFS | up to 6 years
  Progression-free survival (PFS), assessed by investigators (RECIST v1.1)
DoR | up to 6 years
  Duration of response (DoR), assessed by BICR and investigators
DCR | up to 6 years
  Disease control rate (DCR), assessed by BICR and investigators
OS | up to 6 years
  overall survival (OS)
Safety (AE) | up to 6 years
  Incidence and severity of adverse events (AEs)
Number of Participants With Abnormal Laboratory Values or clinical findings | up to 6 years
  Abnormal laboratory or clinical findings
dose-limiting toxicity（DLT） | up to 6 years
  Incidence and severity of dose-limiting toxicity（DLT）
blood concentrations of JS212, JS207,toriplimab, or JS213 | up to 2 years
  Evaluation of blood concentrations of JS212, JS207,toriplimab, or JS213
ADA incidence | up to 4 years
  Incidence and titers of anti-drug antibodies (ADA) for JS212,JS207,toriplimab, or JS213; neutralizing antibodies (NAb) if applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No